CLINICAL TRIAL: NCT02886533
Title: Major Bleeding Risk Associated With Antithrombotics : The SACHA (Surveillance Des Accidents Hémorragiques Graves Sous Antithrombotiques) Study
Brief Title: Major Bleeding Risk Associated With Antithrombotics
Acronym: SACHA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC12_8986_SACHA
Record Dates: First submitted 2016-08-18; First posted 2016-09-01 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2017-02

CONDITIONS: Major Haemorrhage
Keywords: Major haemorrhage; Oral anticoagulation; Antiplatelet drugs; Gastrointestinal bleeding; Intracranial haemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Antithrombotic — Collection of clinical, biological data

SUMMARY:
Prospective, multicenter, observational study with a three-year inclusion period (from January 1, 2012 to December 31, 2015) and a 6-month follow-up

DETAILED DESCRIPTION:
All adults subjects living in the five well-defined areas affiliated to the French National Health Insurance System and having had at least one reimbursement of any antithrombotic in the 3-year study period are identified by using data from the National Health reimbursement database (Système National d'Information Inter-Régimes de l'Assurance Maladie, SNIIR-AM). SNIIR-AM contains individualized, anonymous and comprehensive data for all health spending reimbursements of affiliated subjects, including basic patient demographic data, medical drugs as well as outpatient medical care, prescribed or performed by health-care professionals from both public and private practices. This allows to calculate a denominator (number of person-years of anti-thrombotic drug exposure).

Crude incidence rates of major bleeding per 100 person-months are calculated in antithrombotic users, anticoagulants and others; stratification on a modified HAS-BLED score allows fair comparison between anti-thrombotic drug classes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with major bleeding event associated with antithrombotic drug
* Patient older than 18 years old
* Information on 1 and 6-month follow-up is given pending non-opposition letter

Exclusion Criteria:

* Patients with major bleeding events associated with antithrombotic during hospitalization
* Patients with intentional overdose with antithrombotic drugs
* Patients with multi-trauma
* Patients living outside the defined influence areas of the five participating cities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with major bleeding events associated with antithrombotic
Sampling Method: Probability Sample
Enrollment: 6484 (Actual)
Dates: Start 2013-01-01; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Quantification of the risk of major bleeding of all classes of antithrombotic drugs, in particular the risk of major bleeding of anticoagulants, vitamin K antagonist (VKA) and direct oral anticoagulants (DOAC), in real clinical practice | 6 months
  Unstable hemodynamic (systolic arterial pressure < 90 mmHg or mean arterial pressure < 65 mm Hg), hemorrhagic shock, uncontrollable bleeding, need for transfusions, need for haemostatic procedure (embolization, endoscopic procedure, surgery), or a life-threatened location of bleeding such as intracranial, intra-spinal, intraocular, retroperitoneal, pericardial, thoracic, intra-articular, intramuscular hematoma with compartment syndrome, acute gastrointestinal bleeding

SECONDARY OUTCOMES:
Number of patients receiving treatment for drug-induced haemorrhage | 6 months
Vital status after major bleeding | 1 month
Vital status after major bleeding | 6 months

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Clinique de l'Anjou, Angers
  - CHU d'Angers, Angers
  - Hôpital Inter-Armées, Brest
  - CHU de Brest, Brest
  - Hôpital Privé Sévigné, Cesson-Sévigné
  - Clinique des Cèdres, Échirolles
  - Groupe Hospitalier Mutualiste, Grenoble
  - CHU de Grenoble, Grenoble
  - CHU de Nantes, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - CHU de Rennes, Rennes
  - Centre Hospitalier Privé, Saint-Grégoire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouget J, Balusson F, Roy PM, Viglino D, Pavageau L, Lacut K, Oger E. Management of epistaxis associated with oral antithrombotic drugs in emergency department and impact on prescription thereafter. Clin Otolaryngol. 2023 May;48(3):457-464. doi: 10.1111/coa.14040. Epub 2023 Feb 28. PMID 36789614
- [Derived] Bouget J, Balusson F, Kerbrat S, Roy PM, Viglino D, Lacut K, Pavageau L, Oger E. Clinical use of low-dose parenteral anticoagulation, incidence of major bleeding and mortality: a multi-centre cohort study using the French national health data system. Eur J Clin Pharmacol. 2022 Jul;78(7):1137-1144. doi: 10.1007/s00228-022-03318-x. Epub 2022 Apr 6. PMID 35385975
- [Derived] Bouget J, Balusson F, Viglino D, Roy PM, Lacut K, Pavageau L, Oger E. Major bleeding risk and mortality associated with antiplatelet drugs in real-world clinical practice. A prospective cohort study. PLoS One. 2020 Aug 7;15(8):e0237022. doi: 10.1371/journal.pone.0237022. eCollection 2020. PMID 32764775
- [Derived] Bouget J, Balusson F, Maignan M, Pavageau L, Roy PM, Lacut K, Scailteux LM, Nowak E, Oger E. Major bleeding risk associated with oral anticoagulant in real clinical practice. A multicentre 3-year period population-based prospective cohort study. Br J Clin Pharmacol. 2020 Dec;86(12):2519-2529. doi: 10.1111/bcp.14362. Epub 2020 Jun 1. PMID 32415705